CLINICAL TRIAL: NCT06952790
Title: Fostering Oral Chemotherapy Understanding and Safety (FOCUS) Qualitative Study: Utilization of an Adherence Application
Brief Title: Fostering Oral Chemotherapy Understanding and Safety (FOCUS) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240618
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EveryDose Mobile Application Group (Experimental): Participants in this group will use the EveryDose mobile application for up to 12 weeks.
  Interventions: Behavioral: EveryDose Mobile Application

INTERVENTIONS:
Behavioral: EveryDose Mobile Application — Participants will use this application every day for up to 10 minutes, for up to 12 weeks. The purpose of the application is to improve medication adherence. Participants will receive an alert to the mobile device while at home to ensure medication was taken, and to serve as a medication log.

SUMMARY:
The purpose of this study is to learn about the experiences of cancer patients during treatment utilizing a mobile app called EveryDose© to track prescribed oral treatment for cancer. Based on these experiences, the study team will decide on expanding this pilot study to evaluate other methods that may prove to be beneficial in supporting cancer patient's ability to take cancer medications as prescribed (another common phrase used for this is adherence to treatment).

ELIGIBILITY:
Inclusion Criteria:

* Any sex/gender Able to provide written informed consent
* Able to read/understand English or Spanish
* Diagnosis of hematologic or solid tumor cancer diagnosis
* Prescribed an oral anti-cancer drug as monotherapy treatment for the first time by their treating oncologist.
* Internet access on a smartphone, tablet, or computer

Exclusion Criteria:

* Less than 18 years of age
* Unable to provide written informed consent
* Unable to read/understand English or Spanish
* History of dementia or major psychiatric disease that would interfere with study participation
* Prior treatment with an oral anti-cancer treatment
* Participating in another clinical trial during the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who agree to use the EveryDose application | up to 12 weeks
  Percentage of patients who agree to use the EveryDose application
EveryDose application adherence measured by percentage | up to 12 weeks
  The percentage of weeks out of 12 week-period that the patient used the App (> 50%)
Medication Adherence measured by dose ratio | up to 12 weeks
  Will be measured by the ratio of doses taken to the doses prescribed over a given time period.

SECONDARY OUTCOMES:
Percentage of patient satisfaction measured by SUS | 12 weeks (post intervention)
  Percentage of patients who are satisfied with the EveryDose© mobile app (at least 80%) via the Systems Usability (SUS) survey by providers and patients. Survey asks patient about their satisfaction with the mobile application. Responses range from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No